CLINICAL TRIAL: NCT03320746
Title: Enhancing Physical Activity and Healthy Aging Among Recent Retirees - Randomized Controlled In-home Physical Activity Trial
Brief Title: Enhancing Physical Activity and Healthy Aging Among Recent Retirees
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other); Juho Vainio Foundation (Other); Ministry of Education and Culture, Finland (Other)
Responsible Party: Principal Investigator, Tuija Leskinen, Dr, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 309526
Record Dates: First submitted 2017-10-11; First posted 2017-10-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Exercise; Aging; Retirement
Keywords: Physical activity; Sedentary time; Intervention; Retiree
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity trackers (Experimental): The participants were requested to wear a commercial wrist-worn activity tracker (Polar Loop 2, Polar, Kempele, Finland) every day and night for 12 months.
  Interventions: Device: Polar Loop 2 activity tracker
- No activity trackers (No Intervention): Control group members were requested to abstain from the use of any type of activity trackers and they were informed that they will receive the activity trackers and guidance for using them after the follow-up.

INTERVENTIONS:
Device: Polar Loop 2 activity tracker — The participants were instructed to aim to reach the daily activity goal, initially set at stage 1 as per the goals set by the trackers' manufacturer. The daily activity goal was based on user's typical daily activities, gender and age. The stage 1 daily activity goal corresponded to ~1h/day of jogging or ~2h/day of walking or ~7h/day household activities or a combination of these activities. The tracker gave an inactivity alert as a vibration and text "it's time to move" on the screen of the tracker if the user has been still for 55 minutes.
  Arms: Activity trackers

SUMMARY:
The purpose of REACT project is to provide cost-effective way to promote physical activity and reduce sedentary time among older adults. This is done by examining the efficacy of activity tracker based intervention on wake-time physical activity, sedentary time, sleep and other health outcomes among recent retirees. REACT study will be the first randomized physical activity trial targeted to time window right after retirement.

ELIGIBILITY:
Inclusion Criteria:

* actual retirement date between Jan 2017 and Dec 2018
* maximum of 12 months from the actual retirement
* capable of doing exercise (able to walk 500 m continuously)
* basic knowledge on how to use computer and Internet access at home

Exclusion Criteria:

* current post-operative state or upcoming surgery within the next 6 months
* malign cancer or recent myocardial infraction

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in wake time physical activity | Primarily change from baseline to 12 months, secondarily change from baseline to 3 months and to 6 months.
  Accelerometer based measurement

SECONDARY OUTCOMES:
Change in wake time sedentary activity | Primarily change from baseline to 12 months, secondarily change from baseline to 3 months and to 6 months.
  Accelerometer based measurement
Change in sleep duration and quality | Primarily change from baseline to 12 months, secondarily change from baseline to 3 months and to 6 months.
  Accelerometer based measurement
Change in metabolic profile | Baseline to 12 months
  Fasting blood sample: lipid profile (total cholesterol, HDL, LDL, triglycerides), fasting plasma glucose, HbA1C, and CRP; blood pressure: systolic and diastolic blood pressure; body composition: fat mass, fat free mass, body weight, waist circumference
Change in activity locations | Baseline to 12 months
  GPS-tracking provides data of the latitude, longitude, and time, i.e. when and where an individual is located.

OTHER OUTCOMES:
Change in self-reported health | Baseline to 12 months
  Range 1 to 5 "good to poor"
Change in self-reported functioning | Baseline to 12 months
  SF-36 physical functioning, 10 items, subscale range 1 to 3 "health limits a lot to health does not limit at all", total score range 0 to 10 "no to severe limitations"
Change in self-reported well-being | Baseline to 12 months
  GHQ-12, total score range 0 to 12 points, ≥4 points indicates of psychological distress
Change in diet | Baseline to 12 months
  Index of Diet Quality (IDQ) score, total score range 0 to 15 points, ≥10 points indicates of healthy diet
Change in self-reported exercise motivation | Baseline to 12 months
  Short version of Recreational Exercise Motivation Measure (REMM), subscale range 1 to 5 "strongly disagree to strongly agree"
Change in sleep difficulties | Baseline to 12 months
  Jenkins sleep problem scale, subscale range 1 to 6 "not at all to almost every night"
Change in physical activity social support | Baseline to 12 months
  Modified Social Support for Exercise Scale, subscale range 1 to 3 "never to often", mean score 1 to 3 "low to high"
Change in measured functioning | Baseline to 12 months
  Number of chair test repetitions

CONTACTS AND LOCATIONS:
Overall Officials: Sari Stenholm, Prof, Principal Investigator — University of Turku; Tuija Leskinen, Dr, Principal Investigator — University of Turku
Locations (1):
- University of Turku /Department of Public Health, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized partial datasets of the REACT trial are available by application with bona fide researchers with an established scientific record and bona fide organizations.
Supporting Information: Analytic Code
Time Frame: 2020-2030
Access Criteria: Anonymized partial datasets of the REACT trial are available by application with bona fide researchers with an established scientific record and bona fide organizations.

REFERENCES:
- [Background] Stenholm S, Pulakka A, Kawachi I, Oksanen T, Halonen JI, Aalto V, Kivimaki M, Vahtera J. Changes in physical activity during transition to retirement: a cohort study. Int J Behav Nutr Phys Act. 2016 Apr 16;13:51. doi: 10.1186/s12966-016-0375-9. PMID 27084334
- [Background] Leskinen T, Pulakka A, Heinonen OJ, Pentti J, Kivimaki M, Vahtera J, Stenholm S. Changes in non-occupational sedentary behaviours across the retirement transition: the Finnish Retirement and Aging (FIREA) study. J Epidemiol Community Health. 2018 Aug;72(8):695-701. doi: 10.1136/jech-2017-209958. Epub 2018 Apr 10. PMID 29636399
- [Background] Pulakka A, Leskinen T, Suorsa K, Pentti J, Halonen JI, Vahtera J, Stenholm S. Physical Activity across Retirement Transition by Occupation and Mode of Commute. Med Sci Sports Exerc. 2020 Sep;52(9):1900-1907. doi: 10.1249/MSS.0000000000002326. PMID 32150014
- [Background] Myllyntausta S, Pulakka A, Salo P, Kronholm E, Pentti J, Vahtera J, Stenholm S. Changes in accelerometer-measured sleep during the transition to retirement: the Finnish Retirement and Aging (FIREA) study. Sleep. 2020 Jul 13;43(7):zsz318. doi: 10.1093/sleep/zsz318. PMID 31903480
- [Background] Suorsa K, Pulakka A, Leskinen T, Heinonen I, Heinonen OJ, Pentti J, Vahtera J, Stenholm S. Objectively Measured Sedentary Time Before and After Transition to Retirement: The Finnish Retirement and Aging Study. J Gerontol A Biol Sci Med Sci. 2020 Sep 16;75(9):1737-1743. doi: 10.1093/gerona/glz127. PMID 31095675
- [Background] Myllyntausta S, Stenholm S. Sleep Before and After Retirement. Curr Sleep Med Rep. 2018;4(4):278-283. doi: 10.1007/s40675-018-0132-5. Epub 2018 Oct 24. PMID 30464885
- [Derived] Leskinen T, Suorsa K, Tuominen M, Pulakka A, Pentti J, Loyttyniemi E, Heinonen I, Vahtera J, Stenholm S. The Effect of Consumer-based Activity Tracker Intervention on Physical Activity among Recent Retirees-An RCT Study. Med Sci Sports Exerc. 2021 Aug 1;53(8):1756-1765. doi: 10.1249/MSS.0000000000002627. PMID 34261997
- [Derived] Pasanen S, Halonen JI, Pulakka A, Kestens Y, Thierry B, Brondeel R, Pentti J, Vahtera J, Leskinen T, Stenholm S. Contexts of sedentary time and physical activity among ageing workers and recent retirees: cross-sectional GPS and accelerometer study. BMJ Open. 2021 May 18;11(5):e042600. doi: 10.1136/bmjopen-2020-042600. PMID 34006539
- [Derived] Suorsa K, Leskinen T, Pulakka A, Pentti J, Loyttyniemi E, Heinonen I, Vahtera J, Stenholm S. The Effect of a Consumer-Based Activity Tracker Intervention on Accelerometer-Measured Sedentary Time Among Retirees: A Randomized Controlled REACT Trial. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):579-587. doi: 10.1093/gerona/glab107. PMID 33839766
- See also: Finnish Retirement and Aging Study — http://www.utu.fi/firea